CLINICAL TRIAL: NCT01041716
Title: Clinical and Microbiological Outcomes of Infections Due to Carbapenem-Resistant Gram-Negative Bacteria
Status: Completed | Type: Observational
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09/11VA03
Record Dates: First submitted 2009-12-30; First posted 2010-01-01 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Drug Resistance, Microbial
Keywords: Carbapenem; Klebsiella pneumoniae carbapenemase; Acinetobacter baumannii; Pseudomonas aeruginosa
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: None - Observational study — None - Observational study

SUMMARY:
Carbapenems are a class of antibiotic agents which kill a broad spectrum of bacteria. Infections due to gram-negative bacteria which have acquired resistance to carbapenems are increasing, especially with Klebsiella pneumoniae, Acinetobacter baumannii and Pseudomonas aeruginosa . The optimal treatment of such infections is not known. Antibiotics like polymyxin, tigecycline and rifampin are used alone or in combination with other antibiotics. The outcome of using these new and old drugs is not well studied. This observational study aims to study the clinical and microbiological outcomes of these infections and treatment at our institution.

DETAILED DESCRIPTION:
Objectives

1. To define the demographic and risk factor profile of patients acquiring CRGNB infection.
2. To define the characteristics of CRGNB infection.
3. To report the different treatments employed for CRGNB infection.
4. To report the microbiological and clinical outcomes of different treatment options

   * a. Microbiological outcomes: frequency of microbiological success. Microbiological success will be defined as two successive negative cultures from the same site as from where the CRGNB was originally isolated.
   * b. Clinical outcomes: clinical success (clinical cure), adverse effects of treatment especially the nephrotoxicity in relation to the use of polymyxin, ICU length of stay (if applicable), hospital length of stay, ICU mortality (if applicable), hospital mortality and in-hospital recurrence of infection. Clinical success will be defined as resolution or improvement of clinical symptoms and signs of infection and discontinuation of the antibiotics.

Study duration:

We plan to collect the data for a one year period. Based on the current prevalence rate at our institution, we anticipate having data for 300 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult in-patients (age≥18 years) having an infection due to CRGNB (Klebsiella pneumoniae, Acinetobacter baumannii and Pseudomonas aeruginosa only). CRGNB Infection will be defined as isolation of CRGNB from any source requiring treatment with anti-infective agents with or without manifestations of systemic inflammatory response syndrome.

Exclusion Criteria:

* Patients colonized with CRGNB and not having an active infection.
* Recurrent infection in a previously included patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult in-patients (age≥18 years) having an infection due to CRGNB (Klebsiella pneumoniae, Acinitobacter baumanii and Pseudomonas aeruginosa only). CRGNB Infection will be defined as isolation of CRGNB from any source requiring treatment with anti-infective agents with or without manifestations of systemic inflammatory response syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical success | At the end of treatment
  Resolution (or improvement) of clinical symptoms and signs of infection and discontinuation of the antibiotics.

SECONDARY OUTCOMES:
Microbiological success | At the end of treatment
  Two successive negative cultures from the same site as the original pathogen was isolated.
Recurrence rate | During the hospital stay
  Recurrence of symptoms and signs of infection from the same organism and reinstituion of antibiotic therapy
Adverse effects of treatment | During treatment with antibiotics
  Adverse effects related to antibiotic administration, especially nephrotoxic and neurotoxic effects of polymyxin
Hospital length of stay | During the hospital stay
  Number of days hospitalized
Mortality | During hospital stay
  All cause mortality during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Sriharsha Rao, M.D., Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Bradford PA, Bratu S, Urban C, Visalli M, Mariano N, Landman D, Rahal JJ, Brooks S, Cebular S, Quale J. Emergence of carbapenem-resistant Klebsiella species possessing the class A carbapenem-hydrolyzing KPC-2 and inhibitor-resistant TEM-30 beta-lactamases in New York City. Clin Infect Dis. 2004 Jul 1;39(1):55-60. doi: 10.1086/421495. Epub 2004 Jun 14. PMID 15206053
- [Background] Bratu S, Landman D, Haag R, Recco R, Eramo A, Alam M, Quale J. Rapid spread of carbapenem-resistant Klebsiella pneumoniae in New York City: a new threat to our antibiotic armamentarium. Arch Intern Med. 2005 Jun 27;165(12):1430-5. doi: 10.1001/archinte.165.12.1430. PMID 15983294
- [Background] Patel G, Huprikar S, Factor SH, Jenkins SG, Calfee DP. Outcomes of carbapenem-resistant Klebsiella pneumoniae infection and the impact of antimicrobial and adjunctive therapies. Infect Control Hosp Epidemiol. 2008 Dec;29(12):1099-106. doi: 10.1086/592412. PMID 18973455
- [Background] Weisenberg SA, Morgan DJ, Espinal-Witter R, Larone DH. Clinical outcomes of patients with Klebsiella pneumoniae carbapenemase-producing K. pneumoniae after treatment with imipenem or meropenem. Diagn Microbiol Infect Dis. 2009 Jun;64(2):233-5. doi: 10.1016/j.diagmicrobio.2009.02.004. Epub 2009 Apr 2. PMID 19345034
- [Background] Bratu S, Tolaney P, Karumudi U, Quale J, Mooty M, Nichani S, Landman D. Carbapenemase-producing Klebsiella pneumoniae in Brooklyn, NY: molecular epidemiology and in vitro activity of polymyxin B and other agents. J Antimicrob Chemother. 2005 Jul;56(1):128-32. doi: 10.1093/jac/dki175. Epub 2005 May 25. PMID 15917285